CLINICAL TRIAL: NCT00060411
Title: A Phase I, Pharmacological, and Biological Study of OSI-774 in Combination With FOLFOX 4 (5-FU, Leucovorin, and Oxaliplatin) and Bevacizumab (Avastin) in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03157; NCI-2012-03157 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5869; JHOC-J0220; JHOC-02072506; J0220 02-07-25-06 (Other: Johns Hopkins University); 5869 (Other: CTEP); U01CA070095 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Erlotinib Hydrochloride; Fluorouracil; Leucovorin; Oxaliplatin; Bevacizumab

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive oral elotinib alone once daily for 1 week before the beginning of course 1. Patients then receive oral erlotinib once daily on days 1-28; oxaliplatin IV over 2 hours on day 1; and leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2. Patients also receive bevacizumab IV over 30-90 minutes on day 15 of course 1 and on days 1 and 15 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Biological: bevacizumab

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given IV
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib and bevacizumab with combination chemotherapy may kill more tumor cells. This phase I trial is studying the side effects and best dose of erlotinib when given together with bevacizumab, fluorouracil, leucovorin, and oxaliplatin in treating patients with metastatic or locally advanced colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of OSI-774 given in combination with FOLFOX 4 and Bevacizumab, in patients with advanced colorectal cancer.

II. To characterize the toxicity profile of this regimen. III. To explore the antitumor activity of this combination.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of OSI-774 given with FOLFOX 4, and Bevacizumab.

II. To determine the relationship between CYP3A4 activity and OSI-774 clearance.

III. To correlate Cytochrome P450 activity with OSI-774 PK using midazolam clearance.

IV. To determine the relationship between expression and activation of the EGFR and related signaling pathways and outcome of patients with colorectal cancer patients who are treated with OSI-774 in combination with FOLFOX 4 and Bevacizumab.

V. To explore the biological effects of OSI-774 in patients with advanced colorectal cancer and its relationship with dose and plasma concentration.

VI. To explore the use of fluorodeoxy-glucose (FDG) positron emission tomography (PET) scan to predict the biological effects and outcome of patients with colorectal cancer who are treated with OSI-774 and FOLFOX 4 and Bevacizumab.

VII. To assess 5FU PK when given in this manner, and to correlate with several previously characterized genetic polymorphisms and drug response VIII. To evaluate the association of allelic variants in AAG and OSI-774 disposition.

OUTLINE: This is a dose-escalation study of erlotinib.

Patients receive oral elotinib alone once daily for 1 week before the beginning of course 1. Patients then receive oral erlotinib once daily on days 1-28; oxaliplatin IV over 2 hours on day 1; and leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2. Patients also receive bevacizumab IV over 30-90 minutes on day 15 of course 1 and on days 1 and 15 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 38 patients will be accrued for this study within 19-38 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma with metastatic or locally advanced disease not amenable to curative therapy
* The patients may have therapy for advanced disease completed no less than 28 days prior to enrolling on this protocol; chemotherapy in the adjuvant setting may be allowed, but must have been completed at least 120 days prior to enrollment onto this protocol; prior bevacizumab is allowed
* ECOG performance status =< 1 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin =< 2 mg/dL
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal (=< 5 X institutional upper limit of normal for patients with liver metastatsis)
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* In addition, those patients consenting to have a tumor biopsy and enrolling on that portion of the protocol must have:

  * PTT < 40 seconds
  * PT < 2 seconds more than ULN
* Patients must have unidimensionally-measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Ability to understand and the willingness to sign a written informed consent document
* After the MTD has been defined and 10-20 patients have been treated at this dose level, enrollment will be restricted to patients who have tumor lesions amenable to sequential sampling, if less than 10 patients have had this performed
* Patients undergoing tumor biopsies must not be taking any anti-platelet agents or anticoagulants for at least 5 days prior to biopsy; tumor that will be considered for biopsy will include skin lesions, liver metastases, and peripheral lymph nodes (excluding supraclavicular and high cervical nodes), but will not include lung nodules; if a liver biopsy is being performed, the patient's films (CT or MRI) must be reviewed by the radiologist performing the biopsy (Dr Macura), who must feel that a biopsy is safe and carry minimal risk
* No concurrent nephritic syndrome, uncontrolled hypertension, congestive heart failure

Exclusion Criteria:

* Previous oxaliplatin therapy for metastatic disease; (prior adjuvant therapy with oxaliplatin is allowed as long as 120 days have elapsed since the last oxaliplatin treatment)
* Less than 120 days elapsed time between chemotherapy treatment for adjuvant disease and enrollment onto this protocol or less than 28 days between therapy for metastatic disease and enrollment onto this protocol
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-774, oxaliplatin, 5-FU, or leucovorin
* Patients with a significant neuropathy (greater than grade 2) not controlled despite medications
* Prior treatment with EGFR targeting therapies
* Major surgery or significant traumatic injury occurring within 28 days prior to treatment; all surgical wounds must be healed
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because OSI-774 is an epidermal growth factor inhibitor with the potential for teratogenic or abortifacient effects based on the data suggesting that EGFR expression is important for normal organ development; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-774, breastfeeding should be discontinued if the mother is treated with OSI-774; because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with OSI-774; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients with only non-measurable disease, defined as all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or <10 mm with spiral CT scan) and truly non-measurable lesions, which include the following:

  * Bone lesions;
  * Leptomeningeal disease;
  * Ascites;
  * Pleural/pericardial effusion;
  * Inflammatory breast disease;
  * Lymphangitis cutis/pulmonis;
  * Abdominal masses that are not confirmed and followed by imaging techniques;
  * Cystic lesions
* Patients without sufficient central venous access for therapy
* Patients with thromboembolic events (MI, TIA, stroke, or angina) occurring within the past 6 months prior to the start of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-06; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of OSI-774 given in combination with FOLFOX 4 and Bevacizumab, in patients with advanced colorectal cancer | 28 days
Toxicity profile of this regimen evaluated using the NCI Common Toxicity Criteria Version 2.0 | Up to 4 years
  The frequency of toxicities per organ system and grade will be summarized per each dose level.
Antitumor activity of this combination determined using the RECIST criteria | Up to 4 years
  The percentage of patients in each category of complete response, partial response, stable disease and progressive disease will be calculated using the total number of patients enrolled in an intent to treat analysis.
Overall survival | Up to 12 months
  Will be estimated using the Kaplan-Meier method and will be displayed graphically. Median overall survival and confidence limits will be determined. Kaplan-Meier estimates of survival at 6 and 12 months and their standard errors will be calculated.
Progression-free survival | Up to 12 months
  Progression-free survival will be estimated using the Kaplan-Meier method and will be displayed graphically. Median overall survival and confidence limits will be determined. Kaplan-Meier estimates of survival at 6 and 12 months and their standard errors will be calculated.
The relationship between CYP3A4 activity and OSI-774 clearance | Days -7 to day -1

SECONDARY OUTCOMES:
Pharmacokinetics of OSI-774 given with FOLFOX 4, and Bevacizumab | Days -7 to -1
  Will be determined using conventional non-compartmental and compartmental analysis. The occurrence of pharmacokinetic interactions between oxaliplatin and OSI-774 will be explored by pair comparisons of pharmacokinetic parameters of each agent when given by itself or in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States